CLINICAL TRIAL: NCT01362777
Title: Effects of an In-Patient Individualized Rehabilitation Program on Severity and Symptoms of Obstructive Sleep Apnea Syndrome (OSAS):Results of a Randomized Controlled Pilot Study
Brief Title: Rehabilitation Program as an Alternative Therapy for Moderate to Severe Obstructive Sleep Apnea Syndrome
Acronym: Rehsolvas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: 5 Santé (Other)
Collaborators: A.E.R.O.B.I.E. (Other); INSERM U1046 Physiologie et médecine expérimentale du cœur et des muscles (Unknown)
Responsible Party: Principal Investigator, matthieu.desplan, Docteur M.Desplan (MD), 5 Santé
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF062007
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Sleep Apnea, Obstructive; Metabolic Syndrome
Keywords: Obstructive Sleep Apnea/Hypopnea Syndrome; Exercise training program; Inflammation; Oxidative Stress; Resistance to insulin
MeSH Terms: conditions — Sleep Apnea, Obstructive; Metabolic Syndrome; Inflammation | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- In-Patient Rehabilitation (Experimental): Sessions of rehabilitation contains :
  * Individualized exercise training
  * Educational activities
  * Dietary advices
  Interventions: Behavioral: In-patient rehabilitation
- Educational activities alone (Active Comparator): Out-patient control arm contains only :
  -Educational activities
  Interventions: Behavioral: Educational activities alone

INTERVENTIONS:
Behavioral: In-patient rehabilitation — Individualized exercise training (IET):
  Duration : 24 sessions during 4 weeks
  IET session (2h) contains:
  * 15' start warming up muscles
  * 30' muscle strengthening exercise for arms and abdominal muscles
  * 45' individualized cycle ergometer endurance training to the ventilatory threshold heart rate measured on the cardiopulmonary exercise test.
  * 15' stretching
  * 15' postural, movement and balance exercises IET session was controlled by a professional instructor using heart rate monitoring. Duration, intensity and attendance were recorded in a logbook.
  Educational activities (20h): the 8 themes are comparable to comparator arm. Dietary management: was performed by dietician to ensure that energy intakes are adjusted to energy expenditure. No restrictive diet was prescribe.
  Other Names: Individualized exercise training; Educational activities; Dietary management
  Arms: In-Patient Rehabilitation
Behavioral: Educational activities alone — Educational activities alone contains 10 sessions lasting 1:00 with 8 themes :
  * Physiological mechanisms of apneas/hypopneas
  * Effects of apneas/hypopneas on health (vascular morbidity/mortality and sleepiness)
  * Beneficials effects of CPAP and/or advanced mandibular orthosis
  * Description of sleep stages and physiological roles of sleep
  * Known effects of exercise on sleep and metabolism
  * Importance of good nutritional status and sleep hygiene on quality of life
  * How to apply theses lessons of rehabilitation in daily life
  Other Names: Educational activities
  Arms: Educational activities alone

SUMMARY:
The obstructive sleep apnea/hypopnea syndrome (OSAS) is a common disease (2-4% of the general population) that generates intermittent hypoxemia and sleep fragmentation. OSAS is associated with various metabolic disorders such as metabolic syndrome, type 2 diabetes. OSAS is a risk factor for cardio-vascular diseases by increasing morbidity/mortality. OSAS patients suffer from excessive daytime sleepiness (EDS), a symptom also responsible for at least 30% of traffic accidents but also other cognitive disorders with significant impact on quality of life. OSAS generates oxidative stress, inflammation and resistance to insulin and other systemic metabolic dysregulation of many whose levels are correlated with the severity of the disease.

Treatment with Continuous Positive Airway Pressure (CPAP) has clearly demonstrated its effectiveness to eliminate apneas and improve EDS but it is sometimes difficult to accept and/or poorly tolerated, limiting its effectiveness.

Weight loss and regular physical activity are clearly recommended but rarely done in clinical practice. A few studies have applied to study the effects of rehabilitation training (REE) on the sleep apnea patients and have shown an improvement in sleep quality, reduction of awakenings and arousals from sleep and the Index of Apnea/Hypopnea (AHI), but their methodology was questionable, and the number of patients included was too low.

The investigators hypothesis is that an in-patient multidisciplinary rehabilitation program comprising educational activities, dietary management and individualized exercise training (IET) will decrease OSAS severity, improve sleep quality and symptoms (EDS, fatigue, QoL). This IET program (24 sessions during 4 weeks) could also help to improve many metabolic dysregulation, inflammation and oxidative stress (also markers of cardiovascular risk). Leptin, a hormone involved in regulating appetite, energy expenditure and ventilatory control is increased in OSA (mechanism of leptin resistance). The improved sensitivity to leptin may play a role in enabling a better control of ventilation in these patients.

DETAILED DESCRIPTION:
The obstructive sleep apnea/hypopnea syndrome (OSAS), with an estimated prevalence of between 2 and 4% (1) is characterized by repetitive obstructions of the upper airway that generate intermittent hypoxemia and sleep fragmentation. The typical clinical profile of the apneic patient is an middle aged (50-55 years) obese male, snoring and drowsy. Moreover, OSAS is a risk factor for hypertension independent of obesity (2, 3) and it is now clear evidence that untreated apnea patients have high cardiovascular morbidity / mortality (CVM) higher than subjects treated with CPAP (4-6).

Clinically, excessive daytime sleepiness (EDS) is the main symptom (7) but the attentional and cognitive disorders (8.9), depression or simply a state of fatigue are other possible manifestations of OSAS. The impact on quality of life (QoL) (10-12) are significant and underestimated. The origins of this drowsiness are multiple: one finds the fragmentation of sleep (13,14), intermittent hypoxia, respiratory effort, obesity (15) and certain cytokines such as TNF-alpha and IL-6 involved in sleep regulation (16-19).

On the pathophysiology, the investigators find in the obstructive apneic oxidative stress (20-24) and systemic inflammation (25-27). CRP and levels of some cytokines (IL-1 beta, IL-6, IL-8 and TNF-alpha) are increased and their levels are correlated with the severity of disease as the increase of CVD (28-30 ). Intermittent hypoxia appears to play an essential role in the genesis of these abnormalities (31).

On the metabolic dysregulation of many coexist. Found abnormal fasting blood glucose, a state of insulin resistance, dyslipidemia, and hyperleptinemia. Insulin resistance increases with body weight independent of the index of apnea / hypopnea (AHI) (18, 32-34). Intermittent hypoxia appears to be the cause. Leptin secreted by adipocytes, regulates weight by controlling appetite and energy expenditure. The hyperleptinemia found in OSA is controversial. Obesity appears to be primarily responsible for some (36) while others suggest the role of nocturnal hypoxemia (37). In fact, it is more the state of leptin resistance that hyperleptinemia alone that seems to be involved.

Treatment with continuous positive airway pressure (CPAP) has clearly demonstrated its effectiveness to suppress apneas and sleep fragmentation associated. A meta-analysis (38) has confirmed the improvement of IDS by the PPC. However, in less severe forms, improving the SDE is less clear (39) and the PPC is sometimes not easily accepted, not tolerated and limiting its effectiveness is its poor compliance (40,41). From a pathophysiological point of view, CSF improves systemic inflammation (26,27) and diminishes the CVD (5.6). For cons, the metabolic dysregulation (insulin resistance, hyperleptinemia, dyslipidemia) are improving somewhat CPAP except in patients without obesity (42-44).

The dietary guidelines are essential for the management of this disease is the result for a large part of a healthy lifestyle deleterious. Weight loss, regular physical activity is also clearly recommended but unfortunately rarely performed and / or supported by our healthcare system. Few studies have focused on studying the effects of such treatment on sleep apneic patients. In normal subjects, the effects of exercise on sleep are described in a meta-analysis (45). The practice of regular physical activity endurance improves quality of sleep (45-47). Sleep latency is shorter, there is less change in stages and fewer awakenings and arousals from sleep. Unlike other studies show that in situations where physical activity is reduced (physical inactivity, obesity, or prolonged bed rest, for example) sleep deteriorates, breaks and daytime alertness decreases. The effect of exercise in OSAS (48,49) and especially the training in physical exercise (48) shows an improvement in sleep quality and reduction of awakenings and arousals from sleep and fewer respiratory events (IAH). Pathophysiological point of view, there is a decrease in concentrations of leptin (50-53) and inflammatory cytokines (54-55) in different populations of subjects (healthy, older, obese, or with heart failure). And the investigators know the effects of exercise on carbohydrate metabolism in particular (decreased insulin resistance).

And physical activity improves sleep quality in normal subjects while in parallel it would have an anti-inflammatory. For patients with severe OSAS, our hypothesis is to improve the quality of sleep (SLP rate) and a decrease in AHI and EDS through rehabilitation training (REE) associated with a comprehensive care (patient education, dietary, psychological, ...). On the pathophysiology, this improvement would be through a reduction of biological abnormalities associated with OSA are also markers of cardiovascular risk. Mainly metabolic disorders, oxidative stress and systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Obstructive Sleep Apnea Hypopnea Syndrome (AHI > 15/h)
* Sedentary patient (Activity Voorrips Questionnary score < 9,4)

Exclusion Criteria:

* OSAS already treated by CPAP or other therapy (OAM,...)
* BMI > 40/m²
* Hypnotic and sedative medications
* Cranio-facial malformation
* Obstructive respiratory disease (COPD, asthma,...)
* Instable heart ischemic disease and all

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-11; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Delta of the Apnea/Hypopnea Index (AHI)between the two arms | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Comparing Delta of AHI 4 weeks (J0/J28) after starting the intervention (assessed by polysomnography at inclusion - end monitoring) between the two arms using the Student t test or Wilcoxon test if the distribution is not Gaussian.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu DESPLAN, MD, Principal Investigator — CHU Montpellier, INSERM U1046
Locations (1):
- Clinique du souffle "La Solane", Osséja, France

REFERENCES:
- [Derived] Desplan M, Mercier J, Sabate M, Ninot G, Prefaut C, Dauvilliers Y. A comprehensive rehabilitation program improves disease severity in patients with obstructive sleep apnea syndrome: a pilot randomized controlled study. Sleep Med. 2014 Aug;15(8):906-12. doi: 10.1016/j.sleep.2013.09.023. Epub 2014 Apr 1. PMID 24947878